CLINICAL TRIAL: NCT06530173
Title: Relationship Between Striae Gravidarum and Low-Back Pain Among Pregnant Women: a Cross-Sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ereen Samir Roshdy poules, Ereen Samir Roshdy, Assiut University
Other Study IDs: Striae and Low-Back pain
Record Dates: First submitted 2024-07-27; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain
Keywords: low back pain in pregnancy; stria gravidraum
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
• To improve the quality of pregnant women's lives and provide better control for pregnancy-associated symptoms.

DETAILED DESCRIPTION:
Women commonly experience low back pain (LBP) during pregnancy, and its severity tends to increase as the pregnancy advances. The reported prevalence of LBP among pregnant women varies widely within the literature, ranging from 20% up to 90%(Katonis et al., 2011; Liddle & Pennick, 2015). This is mostly owing to the different definitions and diagnostic criteria of LBP and thus, its real prevalence is still undetermined. In Africa, LBP was found to affect around 50% of pregnant women(Jimoh et al., 2013; Oyeyemi et al., 2013); however and to our knowledge, the prevalence of this condition in Egypt has not been previously described.

Although the occurrence of LBP in pregnancy is typical and would spontaneously resolve after delivery; yet, LBP can be severe enough to negatively impact the quality of pregnant women's lives and increase the health cost burden on them and on the community as well(Kokanali & Caglar, 2019). Furthermore,such a condition can affect women's ability to effectively fulfill their work duties and increase the work loss due to them taking sick leaves or even quitting their jobs(Sencan et al., 2018). Therefore, it is very essential to make every effort not only to reduce such pain, but also to identify itsetiology in order to prevent its occurrence. Although smoking, high body mass index (BMI) and increased workload have been found to be associated with LBP; however, the exact cause of LBP remains unclear(Katonis et al., 2011; Liddle & Pennick, 2015; Sabino & Grauer, 2008).

On the other hand, striaegravidarum (SG) is another common condition found in pregnancy, affecting 55-90% of pregnant women. SG is typically found after the 24th week of gestation as atrophic linear scars on the breasts, abdomen, buttocks, hips, and thighs (Chang et al., 2004; Farahnik et al., 2017). These lesions can cause serious cosmetic problems and pose a psychological burden on pregnant women (Korgavkar & Wang, 2015). Similarly to LBP, the underlying etiology of such a condition is stillunknown. Yet, some have identified several factors that increase its risk, such as young age, large fetus, increased weight gain and high BMI (Farahnik et al., 2017; Korgavkar & Wang, 2015; Picard et al., 2015).

Interestingly, some have suggested thatan interaction between hormonal and mechanical factors as the underlying mechanismof SG formation. At first, the hormonal changes associated with pregnancy may weaken the connective tissue in the skin. Then, as the pregnancy progresses, the resulting mechanical stretching may add to this weakening and result inSG(Farahnik et al., 2017; Korgavkar & Wang, 2015). In a similar manner, the weakening of the connective tissue can affect the spine stability and thus, back pain starts to develop as the mechanical load related to pregnancy increases on the spine (Casagrande et al., 2015).

With that being said, an association between SG and LBP in pregnancy has been recently suggested in a Turkish study byKokanali & Caglar (2019). They found that the presence of SG was more common and its severity was greater among pregnant women with LBP than among those without LBP. They also reported a positive correlation between SG and LBP severity.However, such an association has not been previously investigated among Egyptian women, and therefore, we will conduct this study in order to assessthe association between SG and LBP among pregnant women living in assuit, Egypt

ELIGIBILITY:
Inclusion Criteria:

* • Adult (>18 years) primigravida at 36-37 weeks of gestation. Uncomplicated singleton pregnancy.

Exclusion Criteria:

* • Women with multiple pregnancies.

  * Women having any signs of labor; including detected uterine contractions, rupture of membranes, or cervical dilatation.
  * Women with any systemic disease, such as gestational diabetes or preeclampsia.
  * Women using any medications during pregnancy, except for iron and vitamins supplements.
  * Women using preventive topical treatment for striaegravidarum.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: All healthy pregnant women presenting to the Antenatal care clinic for routine antenatal care visits will be subjected to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Relationship Between Striae Gravidarum and Low-Back Pain Among Pregnant Women | Baseline
  • To assess the association between the presence and severity of striaegravidarum and low back pain among pregnant women

SECONDARY OUTCOMES:
• To determine the prevalence of low back pain among pregnant women. | Baseline
  • To evaluate the effect of women's socio-demographic characteristics on the presence of striae gravidarum or low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sayed Mostafa, Prof, Study Chair; Ahmed Abbas, Associate Prof, Study Director; Mohamed Shahat, Lecturer, Study Director